CLINICAL TRIAL: NCT04499989
Title: Clinical Outcomes of Vaginal Isonicotinic Acid Hydrazide (INH) Administration Prior to T380A Intrauterine Device Insertion in Women Delivered Only by Cesarean Delivery: a Randomized Double Blinded Clinical Trial
Brief Title: Vaginal Isonicotinic Acid Hydrazide (INH) Administration Prior to T380A Intrauterine Device Insertion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, hany farouk, A Professor, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: aswu/353/4/19
Record Dates: First submitted 2020-08-02; First posted 2020-08-05 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: IUCD Complication
MeSH Terms: interventions — Isoniazid

STUDY DESIGN:
Intervention Model Description: double blind randomized trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blind randomized trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- INH (Experimental): 3 vaginal tablet of isonicotinic acid hydrazide self-inserted by the patient 12 hours before IUD insertion.
  Interventions: Drug: INH
- Placebo Comparator (Placebo Comparator): 3 vaginal tablet of Placebo Comparator self-inserted by the patient 12 hours before IUD insertion.
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: INH — 3 vaginal tablet of isonicotinic acid hydrazide self inserted 12 hours before IUD insertion.
  Other Names: isonicotinic acid hydrazide
  Arms: INH
Drug: Placebo Comparator — 3 vaginal tablet of Placebo Comparator self inserted 12 hours before IUD insertion
  Arms: Placebo Comparator

SUMMARY:
To investigate whether vaginal isonicotinic acid hydrazide administered before intrauterine device (IUD) insertion reduces failed insertions, insertion-related complications and pain in in Women Delivered Only by Cesarean Delivery.

DETAILED DESCRIPTION:
Women may experience pain and technical difficulties may be encountered when insertion of an intrauterine device is attempted through a narrow cervical canal. intrauterine device insertion- related complications and side effects are more common among women who had never delivered vaginally.

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant women
* Women that did not receive any analgesics or Dinoprostone in the 24 hours prior to insertion
* Women who delivered only by cesarean section

Exclusion Criteria:

* Women with any uterine abnormalities as congenital anomalies, endometrial lesions, adenomyosis, fibroids.
* Those with a Category 3 or 4 conditions for intrauterine device insertion according to the WHO Medical Eligibility Criteria for contraceptive use
* Allergy to isonicotinic acid hydrazide .
* Women refuse to participate in the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women Delivered Only by Elective Cesarean Section
Enrollment: 220 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
the difference in the pain intensity scores between the study groups | 10 minutes
  the difference in the pain intensity scores between the study groups at IUD insertion BY10 cm visual analog scale score where 0 denotes no pain and 10 denotes the most imaginable pain

SECONDARY OUTCOMES:
Provider ease of insertion | 10 minutes
  Provider ease of insertion was evaluated using a visual analog scale from 0 to 10 cm where 0 denotes very easy insertion and 10 denotes a very difficult insertion.
insertion time | 10 minutes
  IUD insertion time from speculum in to speculum out

CONTACTS AND LOCATIONS:
Overall Officials: nahla w Shady, md, Study Chair — Aswan universirty
Locations (1):
- Aswan University Hospital, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: No